CLINICAL TRIAL: NCT07120282
Title: A Randomized, Multicenter, Phase 2 Study to Evaluate the Efficacy and Safety of Adjuvant Tislelizumab in High-Risk Stage I NSCLC
Brief Title: Study to Evaluate the Efficacy and Safety of Adjuvant Tislelizumab in High-Risk Stage I NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhijie Wang, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5190; ChiCTR2500103192 (Registry Identifier: A Phase 2 Study to Evaluate the Efficacy and Safety of Adjuvant Tislelizumab in High-Risk Stage I NSCLC)
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; 6-pyruvoyltetrahydropterin synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Tislelizumab 400 mg iv, q6w, for up to 1 year; patients are permitted to receive concurrent adjuvant platinum-based doublet chemotherapy (q3w, up to 4 cycles) starting from the first dose of tislelizumab; during concurrent chemotherapy, a tislelizumab dosage of 200 mg iv, q3w is allowed.
  Interventions: Drug: Tislelizumab 400 mg iv, q6w, for up to 1 year for pts in intervention group
- Control group (No Intervention): Patients are permitted to receive postoperative adjuvant platinum - based doublet chemotherapy (q3w, up to 4 cycles).

INTERVENTIONS:
Drug: Tislelizumab 400 mg iv, q6w, for up to 1 year for pts in intervention group — Tislelizumab 400 mg iv, q6w, for up to 1 year; patients are permitted to receive concurrent adjuvant platinum-based doublet chemotherapy (q3w, up to 4 cycles) starting from the first dose of tislelizumab; during concurrent chemotherapy, a tislelizumab dosage of 200 mg iv, q3w is allowed.
  Arms: Intervention group

SUMMARY:
A Randomized, Multicenter, Phase 2 Study to Evaluate the Efficacy and Safety of Adjuvant Tislelizumab in High-Risk Stage I NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent form (ICF) and agree to follow study requirements and assessment schedule.
* Aged 18 years or older.
* Histologically confirmed stage I non - small cell lung cancer (AJCC 9th edition), with tumor size 2cm <= T <=4cm.
* Postoperative pathological report shows at least one high-risk factor (visceral pleural invasion, lymphovascular invasion, STAS, poorly differentiated status, high-grade invasive adenocarcinoma (any structure + high grade structure >=20%, including solid, micropapillary, or complex glands)).
* ECOG performance status 0 or 1.
* PD-L1 expression >=1%.
* No EGFR/ALK sensitive mutations.
* Achieved complete resection (R0) .
* Within 8 weeks after surgery, with full recovery from operation.
* Adequate organ function.

Exclusion Criteria:

* Any previous treatment for current lung cancer, including radiotherapy and systemic anti-tumour therapies (chemotherapy, immunotherapy, targeted therapy, anti-angiogenesis therapy, etc.).
* Prior chest radiotherapy (including lung, oesophageal, mediastinal, or breast cancer).
* Patients with large - cell neuroendocrine carcinoma (LCNEC) or mixed - subtype non - small - cell lung cancer with small - cell components.
* With EGFR/ALK sensitive mutations.
* Underwent segmentectomy or wedge resection only.
* Tumours involving main bronchi, or with obstructive pneumonia/atelectasis (partial or whole lung).
* Active autoimmune disease or history of relapsing autoimmune disease.
* History of interstitial lung disease, drug-induced interstitial lung disease, or radiation pneumonitis needing hormone therapy, or current active interstitial lung disease, or on relevant treatment/intervention.
* Any condition needing systemic corticosteroid (> 10 mg/d prednisone or equivalent) or other immunosuppressant within 14 days before randomisation
* Used other approved systemic immunomodulators (interferon, interleukin - 2, tumour necrosis factor, thymopentin, thymosin α1, etc.) within 4 weeks before first dose.
* Herbs used for cancer control within 14 days before first study
* Live/attenuated vaccine receipt within 4 weeks before enrollment, or plan to receive during study or within 5 months after last tislelizumab dose.
* History of significant disease or conditions affecting organ/system function, per investigator's judgment.
* Severe chronic/active infection needing systemic antibacterial, antifungal, or antiviral therapy (e.g., tuberculosis) within 14 days before first study-drug dose. ·Known HIV infection.
* Allogeneic stem - cell/organ transplant history.
* Active malignancy within 2 years before enrollment, except the specific cancer studied and locally recurrent cancers cured (e.g., excised basal/squamous - cell skin cancer, superficial bladder cancer, cervical/ breast carcinoma in situ).
* Specific conditions and/or alcohol/drug abuse or dependence that may hinder drug administration, affect outcome interpretation, or increase complication risks.
* Pregnant/breastfeeding women, or men/women planning to conceive during the study.
* Participation in another interventional clinical study (except observational studies or follow-up phases).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2029-08-15 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
2 year disease-free survival rate, 2y-DFS rate | From the start of randomization to two years later

SECONDARY OUTCOMES:
disease-free survival, DFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
overall survival, OS | From date of randomization until the date of death from any cause, assessed up to 60 months
Number of Participants with Adverse Events as Assessed by CTCAE v5.0 | From enrollment to the end of systemic anti-tumor treatment at 30 days (90 days for recording irAE )

IPD SHARING:
Plan to Share IPD: No